

#### Statistical Analysis Plan

NCT Number: NCT02415712

Title: Drug Use Surveillance of Fomepizole Intravenous Infusion "Takeda" (All-Case

Surveillance)

Study Number: Fomepizole-5001

Document Version and Date: Version 2.1/01-Aug-2022

Certain information within this document has been redacted (ie, specific content is masked irreversibly from view) to protect either personally identifiable information or company confidential information.

Note; This document was translated into English as the language on original version was Japanese.

### STATISTICAL ANALYSIS PLAN

PRODUCT NAME: fomepizole

S T U D Y T I T L E : Drug Use Surveillance of Fomepizole Intravenous Infusion

PROTOCOL NUMBER :Fomepizole-5001

S P O N S O R : Takeda Pharmaceutical Company Limited



#### TABLE OF CONTENTS

| LIST OF TERMS AND ABBREVIATIONS | 3 |
|---|---|
| ANALYSIS SETS | 6 |
| IMPORTANT IDENTIFIED RISKS, IMPORTANT POTENTIAL RISKS AND IMPORTANT | 6<br>7 |
| MISSING INFORMATION | 7 |
| HANDLING OF TIME WINDOWS | 8 |
| OTHER DATA HANDLING METHODS | 10 |
| HANDLING OF TIME WINDOWS OTHER DATA HANDLING METHODS 1 NUMBER OF SURVEILLANCE SITES & ENROLLED PATIENTS AND PATIENT | Ø |
| DISPOSITION | 12 |
| 1.1 Breakdown of Patients (Patient Disposition) | 12 |
| DISPOSITION | 14 |
| 2.1 Patient Demographics and Baseline Characteristics | 14 |
| 3 TREATMENT DETAILS | 16 |
| 3.1 Administration of Fomepizole IV | 16 |
| 3.2 Interventions/Procedures (Other Than Pharmacotherapy) | 16 |
| 3.3 Administration of Medications (Other than Fomepizole IV) | 16 |
| 4 SAFETY ANALYSES | 18 |
| 4.1 Incidences of Adverse Events and Adverse Drug Reactions/Infections | |
| 4.1.1 Incidences of Adverse Events | 18 |
| 4.1.2 Incidences of Adverse Drug Reactions/Infections | 18 |
| 4.1.3 Incidences of Adverse Events and Adverse Drug Reactions/Infections Identified in | |
| the Safety Specification | 19 |
| 4.2 Incidences of Adverse Events and Adverse Drug Reactions/Infections in Patients | |
| Excluded from the Safety Analysis Set | 20 |
| 4.2.1 Incidences of Adverse Events in Patients Excluded from the Safety Analysis Set | 20 |
| 4.2.2 Incidences of Adverse Drug Reactions/Infections in Patients Excluded from the | |
| Safety Analysis Set | 21 |
| 4.3 Incidences of Adverse Events and Adverse Drug Reactions/Infections by Seriousness, | |
| Time of Onset, Outcome, and Causal Relationship with Fomepizole IV | 21 |
| 4.3.1 Incidences of Adverse Events by Seriousness, Time of Onset, Outcome, and Causal | |
| Relationship with Fomepizole IV | 21 |
| 4.3.2 Incidences of Adverse Drug Reactions/Infections By Seriousness, Time of Onset, | |
| and Outcome | 22 |
| 4.4 Incidences of Serious Adverse Events and Adverse Drug Reactions/Infections | 22 |
| 4.4.1 Incidences of Serious Adverse Events | 22 |
| 4.4.2 Incidences of Serious Adverse Drug Reactions/Infections | 23 |

| 4.5 Factors Potentially | Affecting Safety | |
|---|---|---|
| 4.5.1 Incidences of | Adverse Drug Reactions/Infections by Patient Demographics & | |
| Baseline Char | racteristics and Treatment Details23 | orms of |
| 4.5.2 Incidences of | Adverse Drug Reactions/Infections by Seriousness, Deaths, Patient | ۱. |
| Demographic | s & Baseline Characteristics and Treatment Details24 | O) |
| 4.5.3 Incidences of | Adverse Drug Reactions/Infections by Sex | ins |
| 4.5.4 Incidences of | Adverse Drug Reactions/Infections by Age Bracket25 | SI |
| | Adverse Drug Reactions/Infections by Alcohol Consumption (Y/N)25 | |
| 4.5.6 Incidences of | Adverse Drug Reactions/Infections by Administration of Fomepizole | |
| IV | 26 | |
| | Adverse Drug Reactions/Infections by Intervention/Procedure (Other | |
| than Pharmac | otherapy) 26 | |
| | Adverse Drug Reactions/Infections by Administration of Medications | |
| (Other than Fo | omepizole IV)26 | |
| 4.5.9 Incidences of | Adverse Drug Reactions/Infections by Presence or Absence (Y/N) of | |
| Toxic Sympto | oms | |
| 4.6 Time Courses of T | bms | |
| 4.6.1 Time Courses | of Vital Signs27 | |
| 4.6.2 Time Courses | of Laboratory Test Parameters | |
| 5 EFFICACY ANALYSE | ES | |
| 5.1 Time Course of Ar | terial Blood pH29 | |
| 5.2 Time Courses of P | oisoning/Toxicity Test Parameters | |
| 5.3 Time Courses of T | Foxic Symptoms | |
| 5.4 Outcome | 31 | |
| 5.5 Factors Potentially | Affecting Efficacy | |
| 6 INCIDENCE OF ADV | ERSE DRUG REACTIONS/INFECTIONS IN THE | |
| SUPPLEMENTARY P | HARMACOVIGILANCE PLAN | |
| 6.1 Incidence of Adve | rse Drug Reactions/Infections in the Supplementary | |
| Pharmacovigilan | ce Plan (Attached Form 12) | |
| 7 SUMMARY OF PATIE | ENTS IN POSTMARKETING SURVEILLANCE34 | |
| 7.1 Summary of Patien | nts in Postmarketing Surveillance (Attached Form 16)34 | |
| 7.1 Summary of Patien Document History (Version [Attachment 1] Amendmen | n Control) | |
| [Attachment 1] Amendmen | nt Comparison Table1 | |
| 200 | | |

#### LIST OF TERMS AND ABBREVIATIONS

- Fomepizole IV: The study drug Fomepizole Intravenous Infusion "Takeda" shall be abbreviated as "fomepizole IV"
- AE: Adverse event occurring after administration of fomepizole IV
- ADRs, etc.: An abbreviation for "adverse drug reactions/infections" that refers to AEs other than
  those with a causal relationship to fomepizole IV as assessed by the investigator as "not related."
  In this SAP, the term is denoted using the full wording "Adverse Drug Reactions/Infections" in
  titles and is abbreviated as "ADRs, etc." in the text and tables.
- SAE: Adverse event assessed as "serious" by the investigator. Any event listed in the MedDRA code list (PT code) of the Important Medical Events List provided under the title "Takeda Medically Significant AE List" is to be handled as serious even if said event was assessed by the investigator as "not serious."
- "Related": AEs with a causal relationship with fomepizole IV that is assessed as either "related"
  or "not evaluable" by the investigator will be handled as "related" AEs.
- Summary statistics: A term that collectively refers to the number of patients, mean value, standard deviation, maximum value, minimum value, and quartile value.
- Number of days after fomepizole IV dosing: The day before the start of fomepizole IV dosing is referred to as Day -1, while the day on which fomepizole IV dosing is commenced is referred to as Day 1.
- Duration of fomepizole IV treatment (days): Final day of fomepizole IV dosing start date of fomepizole IV dosing + 1
- Time & date of completion of fomepizole IV treatment: The time and date at completion of the final infusion of fomepizole IV as recorded in the CRF.
- Patients with faxed Contact Forms: Refers to the patients for whom a completed Contact Form
  has been transmitted by fax and received by the Central Enrollment Center.
- Enrolled patients: Patients whose enrollment was approved by the PMS system.
- Unenrolled patients: Patients with faxed/received Contact Forms whom the PMS system has not approved for enrollment.
- Patients without submitted CRFs: Refers to enrolled patients for whom a CRF has not been submitted/collected.
- Patients with submitted CRFs: Refers to enrolled patients for whom a CRF has been submitted/collected.

- Time of onset of AEs (or ADRs, etc.): Calculated by subtracting the start date of fomepizole IV treatment from the date of onset of the AE (or ADR, etc.) and adding 1 (i.e., adding 1 day).
- Patients with concurrent diabetes mellitus: Patients for whom the box for "Diabetes mellitus" in
  the "Concurrent (coexisting) disease" section of the CRF has been checked. Or other disease:
  Refers to patients with a concurrent disease recorded in the disease name field of the CRF that
  corresponds to standardized MedDRA query (herein "SMQ") code 20000041
  (Hyperglycaemia/new onset diabetes mellitus SMQ [scope: narrow]).
- Patients with concurrent hypertension: Patients for whom the box for "Hypertension" in the
  "Concurrent (coexisting) disease" section of the CRF has been checked. Or other disease: Refers
  to patients with a concurrent disease recorded in the disease name field of the CRF that
  corresponds to SMQ code 20000147 (Hypertension SMQ [scope: narrow]).
- Patients with concurrent dyslipidaemia: Patients for whom the box for "Dyslipidaemia" in the
  "Concurrent (coexisting) disease" section of the CRF has been checked. Or other disease: Refers
  to patients with a concurrent disease recorded in the disease name field of the CRF that
  corresponds to SMQ code 20000026 (Dyslipidaemia SMQ [scope: narrow]).
- Patients with concurrent hyperuricaemia: Patients for whom the box for "Hyperuricaemia" in the
  "Concurrent (coexisting) disease" section of the CRF has been checked. Or other disease: Refers
  to patients with a concurrent disease recorded in the disease name field of the CRF that
  corresponds to MedDRA PT code 10020903 (Hyperuricaemia).
- Patients with concurrent liver disorder: Patients for whom any of the boxes for "Fatty liver,"
   "Alcoholic hepatitis," "Chronic hepatitis," or "liver cirrhosis" in the "Concurrent (coexisting) disease" section of the CRF has been checked. Or other disease: Refers to patients with a concurrent disease recorded in the disease name field of the CRF that corresponds to SMQ code 20000005 (Hepatic disorders SMQ [scope: narrow]).
- Patients with concurrent renal disorder: Patients for whom the box for "Chronic renal disorder" in the "Concurrent (coexisting) disease" section of the CRF has been checked. Or other disease:
   Refers to patients with a concurrent disease recorded in the disease name field of the CRF that corresponds to the Takeda MedDRA query (herein "TMQ") (Renal Disease) or TMQ (Renal Impairment).
- Patients with other concurrent diseases: Patients whose concurrent disease does not fall under the
  above-listed categories of (i.e., concurrent diabetes mellitus, concurrent hypertension, concurrent
  dyslipidaemia, concurrent hyperuricaemia, concurrent liver disorder or concurrent renal
  disorder).

- GCS: The sum of Glasgow Coma Scale (GCS) scores will be calculated for 3 items: eye opening (E), best verbal response (V), and best motor response (M).
- 3-3-9 rating system (JCS): When expressing the Japan Coma Scale (JCS) score numerically, the following categories are used.
  - Score of 0 is recorded as "0 (Alert)"
  - Scores of 1, 2 and 3 are recorded as "I"
  - Scores of 10, 20 and 30 are recorded as "II"
  - Scores of 100, 200 and 300 are recorded as "III"
- Time from ingestion of toxic substance to start of fomepizole IV treatment:
  - Calculated by subtracting the time/date of ingestion (confirmed or estimated) recorded in
    the Toxic Symptoms column of the CRF from the time/date of starting treatment with
    fomepizole IV. Estimated times for "time X" will be expressed as X hr:00mins. Any
    missing data for time or date will be handled as "unknown."
- Ethanol: Drugs with a medicinal product code starting with 2615702 or 2615704.
- Vitamin B6 preparations: Drugs with a medicinal product code starting with 3134001, 3134002, 3134003, 3134004, 3134400 or 3134402.
- Vitamin B1 preparations: Drugs with a medicinal product code starting with 3121001 or 3121400.
- Folic acid preparations: Drugs with a medicinal product code starting with 3135.
- Sodium bicarbonate preparations: Drugs with a medicinal product code starting with 2344004,
   2344005 or 3929400.
- Potassium chloride preparations: Drugs with a medicinal product code starting with 3229001, 3229002 or 3229400.

  Potassium chloride preparations: Drugs with a medicinal product code starting with 3229001, 3229002 or 3229400.

#### ANALYSIS SETS

The DUS all-case surveillance was designed with a "Safety Analysis Set" and an "Efficacy Analysis Set." These analysis sets are defined below.

#### Safety Analysis Set

The Safety Analysis Set is defined as "the set of patients who received fomepizole IV, who did not commit any significant breaches of the DUS Protocol, and in whom the safety of fomepizole IV could be evaluated." Patients for whom CRFs were submitted/collected and who met any of the following criteria were excluded from the Safety Analysis Set.

- Patients who did not receive treatment with fomepizole IV
- Patients in whom the presence or absence of AEs could not be determined (i.e., was "unknown")
- Efficacy Analysis Set

The Efficacy Analysis Set is defined as "the Safety Analysis Set patients who did not commit any significant breaches of the DUS Protocol and in whom the efficacy of fomepizole IV could be evaluated." The Efficacy Analysis Set consisted of the patients in the Safety Analysis Set after excluding the following patients.

- Patients who did not meet the indication for treatment with fomepizole IV
- Patients for whom there is no efficacy data: Patients who met all of the following criteria are regarded as having no efficacy data.
  - There is no available data for arterial blood pH at the start of fomepizole IV dosing (i.e., at baseline), and there is no available data for arterial blood pH from at least one assessment timepoint from 30 minutes (herein denoted as "0.5 hr") after starting fomepizole IV dosing up to 24 hours after completing the final fomepizole IV infusion.
- There is no available data for at least one of the poisoning/toxicity test parameters (PaCO<sub>2</sub>, PaO<sub>2</sub>, bicarbonate ion, BE, anion gap, blood ethylene glycol concentration, blood glycolic acid concentration, blood methanol concentration, blood formic acid concentration, and osmotic pressure gap) at baseline, and there is no available data for at least one of these parameters from at least one assessment timepoint from 0.5 hr after starting fomepizole IV dosing up to 24 hours after completing the final infusion.
- There is no available data for at least one toxic symptom parameter at baseline nor at completion of the final fomepizole IV infusion.
- Outcome has not been documented.

#### IMPORTANT IDENTIFIED RISKS, IMPORTANT POTENTIAL RISKS AND IMPORTANT MISSING INFORMATION

- Important Identified Risks
  - Anaphylaxis: Events that fall under the MedDRA PT codes 10002198 (anaphylactic reaction), 10002199 (anaphylactic shock), 10002216 (anaphylactoid reaction), and 10063119 (anaphylactoid shock).
- Important Potential Risks
- ble terms of Use Central nervous system disorder: An event that meets the MedDRA SOC Code 10029205 (nervous system disorders).
  - Fetal disorder due to drug exposure during pregnancy: An event that corresponds to SMQ Code 20000185 (Pregnancy and neonatal topics) (broad).
- **Important Missing Information**
- Clinical experience in Japanese patients: Events that occurred in patients within Japan. ated anese pat a All patients enrolled in this DUS are located within Japan and are therefore within the scope of "Clinical experience in Japanese patients" so no additional tabulations will be

#### HANDLING OF TIME WINDOWS

Evaluable test parameter data (i.e., data deemed not to be missing any elements and able to be used in the statistical analyses) shall be handled as described below.

Evaluable data that was collected within the relevant time window will be used. If multiple elements of evaluable data exist within the same time window, the data obtained from the test performed closest to the reference time/date will be used. If the time elapsed from the reference time/date is identical or if no reference time/date has been stipulated, the subsequently-obtained data will be used. The amount of time elapsed from the reference time/date shall be determined based on the time elapsed from dosing. If data for the time/date of the test is missing or incomplete, the test timing printed on the CRF shall be used. (As this data is obtained at the time of hospitalization due to poisoning, the integrity/reliability of the test timepoints recorded in the CRF are deemed to be greater than those of other data elements and will therefore be used for the analysis.) If there is a mix of both missing and available data for the time/date of tests at the same assessment timepoint, the data that actually contains the test time/date will be used.

| Test Parameters | for Vital | Signs, L | aboratory ' | Tests and | Toxic Symptoms |
|---|---|---|---|---|---|

| Assessment time | Reference time/date | Time window |
|---|---|---|
| point | Reference time/date | Time after dosing |
| Start of fomepizole IV | treatment -108 hr after start of fom | epizole IV treatment |
| At start of fomepizole IV treatment | At start of fomepizole FV treatment | -48 hr $\leq$ fomepizole IV infusion start time/date $\leq$ 0 hr |
| 0.5 hr after starting<br>fomepizole IV<br>treatment | Fomepizole FV infusion start<br>time/date + 0.5 hr | 0 hr < fomepizole IV infusion start time/date $\leq$ 2 hr |
| 4 hr after starting<br>fomepizole IV<br>treatment | Fomepizole IV infusion start<br>time/date + 4 hr | 2 hr < fomepizole IV infusion start time/date ≤ 6 hr |
| 8 hr after starting fomepizole treatment | Fomepizole IV infusion start<br>time/date + 8 hr | 6 hr < fomepizole IV infusion start time/date $\leq$ 10 hr |
| 12 hr after starting<br>fomepizole IV<br>treatment | Fomepizole IV infusion start<br>time/date + 12 hr | 10 hr < fomepizole IV infusion start time/date $\leq$ 14 hr |
| 16 hr after starting<br>fomepizole IV<br>treatment | Fomepizole IV infusion start<br>time/date + 16 hr | 14 hr < fomepizole IV infusion start time/date $\leq$ 18 hr |
| 20 hr after starting<br>fomepizole IV<br>treatment | Fomepizole IV infusion start<br>time/date + 20 hr | 18 hr < fomepizole IV infusion start time/date $\leq$ 22 hr |
| 24 hr after starting<br>fomepizole IV<br>treatment | Fomepizole IV infusion start<br>time/date + 24 hr | 22 hr < fomepizole IV infusion start time/date ≤ 30 hr |
| 36 hr after starting<br>fomepizole IV<br>treatment | Fomepizole IV infusion start<br>time/date + 36 hr | 30 hr < fomepizole IV infusion start time/date $\leq$ 42 hr |

| Time after dosing V infusion start 42 hr < fomepizole IV infusion start time/date ≤ 54 hr |
|---|
| V influsion start 42 hr < formanizada IV influsion start time/data < 54 hr |
| e + 48 hr |
| V infusion start<br>+ 60 hr 54 hr < fomepizole IV infusion start time/date ≤ 66 hr |
| V infusion start<br>+ 72 hr 66 hr < fomepizole IV infusion start time/date ≤ 78 hr |
| V infusion start<br>+ 84 hr |
| V infusion start<br>+ 96 hr 90 hr < fomepizole IV infusion start time/date ≤ 102<br>hr |
| V infusion start<br>+ 108 hr 102 hr < fomepizole IV infusion start time/date ≤ 114<br>hr |
| urs after end of final infusion of fomepizole IV |
| inal fomepizole IV $0.5 \text{ hr} \le \text{end time/date of final fomepizole IV} $ infusion $\le 6 \text{ hr}$ |
| inal fomepizole IV 6 hr < end time/date of final fomepizole IV infusion ≤ 18 hr |
| inal fomepizole IV 18 hr < end time/date of final fomepizole IV infusion<br>+24 hr ≤ 30 hr |
| 0 hr < fomepizole IV infusion start time/date ≤ 114 hr; or -0.5 hr ≤ end time/date of final fomepizole IV infusion ≤ 30 hr; whichever assessment timepoint is sooner |
| IV te |

#### OTHER DATA HANDLING METHODS

- Displayed decimals/numerical data will be handled according to the following rules.
  - Percentages (%):
- ... Round percentage to the second decimal place and ... To the second decimal place.

  Other data elements: Round percentage to the first decimal place and display up to the first decimal place.

  mary statistics:

  Means: Round ...
  - Summary statistics:
    - Means: Round off raw data in the double digits and display up to single digit.
    - Standard deviations: Round off raw data in the triple digits and display up to double digits.
    - Minimum and maximum values: Display this data using the same method as that for raw data.
    - First quartile, median, third quartile: Display raw data up to single digits.
  - P values: Round down (i.e., truncate) to the third decimal place and display up to the third decimal place. When the P value truncated to the third decimal place is <0.001, display as P<0.001.
- Use a two-sided significance level of 5%.
- Missing data for the date (i.e., day, month and year) of AE onset will be handled as follows.
  - If the day of onset is the only data that is missing, and if the month and year of AE onset is identical to those of the initial fomepizole IV treatment, the day of onset shall be regarded as the day on which fomepizole IV dosing commenced (i.e., the event shall be regarded as having occurred on the day of initial fomepizole IV dosing). In all other situations, the day of onset shall be regarded as the first day (i.e. the 1st) of the month.
    - If data for both the day and month are missing, and if the year of AE onset is identical to that of the initial fomepizole IV treatment, the day of onset shall be regarded as the day on which fomepizole IV dosing commenced (i.e., the event shall be regarded as having occurred on the day of initial fomepizole IV dosing). In all other situations, the day and month of onset shall be regarded as the 1st of January.
  - If data on the day, month and year are all missing, the AE onset date will be regarded as missing data.

Property of Takeda: For non-commercial use only and subject to the applicable Temes of Use • If the same patient has been treated on multiple occasions (e.g., if the patient has attempted

# NUMBER OF SURVEILLANCE SITES & ENROLLED PATIENTS AND PATIENT the applicable reims of Use DISPOSITION

#### 1.1 **Breakdown of Patients (Patient Disposition)**

Analysis set: All-Case (enrolled patients) Data element Number of patients enrolled

analyzed:

Number of sites where patients

are enrolled

Patients for whom CRFs were

not submitted/collected

Patients for whom CRFs were

submitted/collected

Patients excluded from Safety

Analysis Set\*

Patients who did not receive fomepizole IV, Reason for exclusion

patients whom presence or absence of AEs (duplicate count)

is unknown:

Safety Analysis Set

Patients excluded from Efficac

Analysis Set\*

Reason for exclusion [Did not meet fomepizole IV indication, no (duplicate count) efficacy data]

Efficacy Analysis Set

Analysis method:

Property of Lakeda. For

The following analyses will be performed and the Patient Disposition diagram will be prepared for the above-mentioned data elements.

The number of surveillance sites will also be shown for patients for whom the Contact Form was transmitted/received by fax and for enrolled patients. If the surveillance is conducted in different departments at the same site, the site shall be counted only once (i.e., as a single site). If no patients meet the criteria for exclusion, said number of patients shall be listed as "0". The numbers of patients excluded from the Safety Analysis Set and from the Efficacy Analysis Set will be tabulated and listed along with the reasons for exclusion.

\* "Patients excluded from the Safety Analysis Set" refers to the patients for whom CRFs were submitted/collected and were also excluded from the Safety Analysis Set. \* Similarly, "patients excluded from the Efficacy Analysis Set" refers to the patients for whom CRFs were submitted/collected and were also excluded from the Efficacy Analysis Set.

#### Frequency tables

Property of Takeda; For non-commercial use only and subject to the applicable Tames of use

#### PATIENT DEMOGRAPHICS AND BASELINE CHARACTERISTICS

#### **Patient Demographics and Baseline Characteristics** 2.1

Safety Analysis Set Analysis set:

Data element Sex

analyzed:

Age (years)

Livin <= - < 65, 65 <= - <= Max, Unknown]
[Min <= - < 65, 65 <= - <= 74, 75 <= - <= Max, Unknown]
[Min <= - < 20, 20 <= 40 <-

40 <= - <= 49, 50 <= - <= 59, 60 <=

69, 70 <= - <= 79, 80 <= **X** = **Max**,

Unknown]

[Ethylene glycol poisoning, suspected Diagnosis (final diagnosis)

ethylene glycol poisoning, methanol

poisoning, suspected methanol poisoning,

other disease, unknown]

Hypersensitivity [no, yes, unknown]

Concurrent (coexisting) disease [no, yes, unknown]

Details of any concurrent [Diabetes mellitus, hypertension,

(coexisting) disease (duplicate dyslipidaemia, hyperuricaemia, liver

disorder, renal disorder, other]

Previous medical history [no, yes, unknown]

Height (cm)  $|Min| \le - < 150, 150 \le - < 160, 160 \le - <$ 

170, 170 <= - <= Max, Not measured]

Body weight (kg)  $|Min| \le - < 50.0, 50.0 \le - < 60.0, 60.0 \le -$ 

Not measured]

[Min <= - < 18.5, 18.5 <= - < 25.0, 25.0 <= -BMI (kg/m<sup>2</sup>)

 $< 30.0, 30.0 \le - \le Max, Not measured$ 

Alcohol consumption (at time of [no, yes, unknown]

poisoning)

Property of Lakedai. For hot Pregnancy (females only) [no, yes, unknown]

Level of consciousness [GCS, 3-3-9 rating system (JCS), unknown]

(duplicate count)

Level of consciousness details

**GCS** [minor (14/15), moderate (9-13), severe (3-

8)]

3-3-9 rating system (JCS) [0 (alert), I, II, III]

Circumstances of poisoning

Ingested substance (duplicate

count)

Data available on time from

ingestion of toxic substance

to start of fomepizole IV

treatment (Yes/No)

Details of "Yes" for data

available on time from

ingestion of toxic substance

to start of fomepizole IV

[Min <= - < 6, 6 <= - < 12, 12 <= - < 24, 24 <= - <= Max]

ral, inhalation. Route of ingestion

Reason ingested [accidental ingestion, suicide attempt, other,

unknown]

Analysis method: Frequency tables of calculated values and summary statistics of measured values will be prepared for the above-mentioned data elements.

Listings will be prepared for details of concurrent (coexisting) diseases (other Archaested, a gested, a gested, a roperty of takeda. For noncommercial property of takeda. diseases) and circumstances of poisoning (ingested substance and amount, time and date ingested, route of ingestion, reason ingested).

#### 3 TREATMENT DETAILS

#### Administration of Fomepizole IV 3.1

Safety Analysis Set Analysis set:

Data element Initial dose of fomepizole IV (mg)

analyzed:

Fomepizole IV treatment duration

(days)

Fomepizole IV cumulative dose (mg)

 $[1, 2, 3, 4, 5, 6, 7, 8, 9, 10, \ge 11]$   $[Min \le - < 30, 30 \le - < 60, 60 \le 90, 90 \le - < = Max]$ Maximum number of infusions

Mean duration of single infusion

(min)

[15 mg/kg, 10 mg/kg, Other] Infusion dose per body weight [Therapeutic objective achieved, Reason for discontinuation of

fomepizole IV (duplicate count) occurrence of AE, inadequate response,

other

Analysis method: Frequency tables of calculated values and summary statistics of measured values

will be prepared for the above-mentioned data elements.

#### Interventions/Procedures (Other Than Pharmacotherapy) 3.2

Safety Analysis Set Analysis set:

Data element Acute blood purification therapy [no, yes]

Details of any (i.e., "Yes") acute blood analyzed: [continuous renal replacement

purification therapy (duplicate count) therapy, plasma exchange,

adsorption, intermittent renal

replacement therapy, other]

Respiratory management (mechanical [no, yes]

ventilation)

GI decontamination [no, yes]

Details of any (i.e., "Yes") GI [gastrolavage, induced emesis,

decontamination therapy (duplicate other]

count)

Analysis method: Frequency tables will be prepared for the above-mentioned data elements.

#### Administration of Medications (Other than Fomepizole IV)

Analysis set: Safety Analysis Set Data element Administration of medication (other than [no, yes]

analyzed: fomepizole IV)

Details of administered medication (other

than fomepizole IV)

Medication name (duplicate count) [ethanol, vitamin B6, vitamin B1,

folic acid preparations, sodium

bicarbonate preparations,

potassium chloride

preparations, others]

No. of medications used

Reason for use (duplicate count) [treatment of AE, treatment of

concurrent (coexisting)

disease, treatment of

underlying disease

(poisoning), other

(prophylaxis, etc.)]

Analysis method: Frequency tables of calculated values and summary statistics of measured values able amber of amber of the contract of the con will be prepared for the above-mentioned data elements. Reason for use will be

calculated by the number of occasions used and number of patients treated.

#### SAFETY ANALYSES

#### Incidences of Adverse Events and Adverse Drug Reactions/Infections 4.1

#### 4.1.1 Incidences of Adverse Events

Analysis set: Safety Analysis Set

Data element **AEs** 

analyzed:

Analysis method: AEs will be analyzed as follows.

- No. of patients with AEs (1)
- (2) No. of AEs
- (3) Incidence rate of AEs
- (4) AE category

Each of these data elements will be determined as follows.

No. of patients with AEs:

The number of patients who develop an AE

No. of AEs:

The number of AEs that occur. If the same AE occurs multiple times in the same patient, the total number of occurrences will be tabulated.

Incidence rate of AEs:

Calculated as follows: No. of patients with AE ÷ No. of patients in the Safety Analysis Set × 100

AE category:

- AEs will be coded using the MedDRA/J terms. AEs will be broadly classified into SOC and tabulated according to PT. AEs belonging to the SOC "Investigations" will be tabulated by HLGT (listed in ascending order of HLGT code but not output) and PT.
  - At the SOC level, the numbers and incidence rates of AEs will be described according to the internationally-recognized SOC order. Patients with multiple occurrences of the same SOC will be counted as a single patient within said SOC.
- At the PT level, the numbers and incidence rates of AEs will be described according to the PT code ascending order. Patients with multiple occurrences of the same PT will be counted as a single patient within said PT.

# Property of Takedai. For not 4.1.2 Incidences of Adverse Drug Reactions/Infections

Analysis set: Safety Analysis Set Data element

ADRs, etc.

analyzed:

Analysis method:

AEs will be analyzed as follows.

- (1) No. of patients with ADRs, etc.
- (2) No. of occurrences of ADRs, etc.
- (3) Incidence rate of ADRs, etc.
- (4) Category of ADRs, etc.

Each of these data elements will be determined as follows.

No. of patients with ADRs, etc.:

• The number of patients who develop ADRs, etc.

Number of occurrences of ADRs, etc.:

The number of times that ADRs, etc. occur. If the same ADR, etc. occurs
multiple times in the same patient, the total number of occurrences will be
tabulated.

Incidence rate of ADRs, etc.:

 Calculated as follows: No. of patients with ADRs, etc. ÷ No. of patients in the Safety Analysis Set × 100

Category of ADRs, etc.:

- ADRs, etc. will be coded using the MedDRA/J terms. AEs will be broadly
  classified into SOC and tabulated according to PT. AEs belonging to the
  SOC "Investigations" will be tabulated by HLGT (listed in ascending order
  of HLGT code but not output) and PT.
- At the SOC level, the numbers and incidence rates of ADRs, etc. will be
  described according to the internationally-recognized SOC order. Patients
  with multiple occurrences of the same SOC will be counted as a single
  patient within said SOC.
- At the PT level, the numbers and incidence rates of ADRs, etc. will be
  described according to the PT code ascending order. Patients with multiple
  occurrences of the same PT will be counted as a single patient within said
  PT.
- 4.1.3 Incidences of Adverse Events and Adverse Drug Reactions/Infections Identified in the Safety Specification
- 4.1.3.1 Incidences of Adverse Events Identified in the Safety Specification (Tabulated By Risk)

Analysis set:

Safety Analysis Set

Data element AEs identified in the Safety Specification (important identified risks and

analyzed: important potential risks)

Stratification Seriousness [serious, not serious]

variable:

Analysis method: The above-mentioned data elements will be analyzed by risk using the same

method described in section 4.1.1 for each stratum of the stratification variables.

Patients with multiple occurrences of the same SOC/PT will be counted as a

single patient within said SOC/PT. However, patients who experience multiple

AEs of varying seriousness will be separately counted as a single patient for the serious event and the non-serious event. Risks to be analyzed shall adhere to the

definitions outlined in the Important Identified Risks, Important Potential Risks,

and Important Missing Information.

## 4.1.3.2 Incidences of Adverse Drug Reactions/Infections Identified in the Safety Specification (Tabulated By Risk)

Analysis set: Safety Analysis Set

Data element ADRs, etc. in the Safety Specification (important identified risks and important

analyzed: potential risks)

Stratification Seriousness [serious, not serious]

variable:

Analysis method: The above-mentioned data elements will be analyzed by risk using the same

method described in section 4.1.2 for each stratum of the stratification variables.

Patients with multiple occurrences of the same SOC/PT will be counted as a

single patient within said SOC/PT. However, patients who experience multiple

AEs of varying seriousness will be separately counted as a single patient for the

serious event and the non-serious event. Risks to be analyzed shall adhere to the

definitions outlined in the Important Identified Risks, Important Potential Risks,

and Important Missing Information.

## 4.2 Incidences of Adverse Events and Adverse Drug Reactions/Infections in Patients Excluded from the Safety Analysis Set

#### 4.2.1 Incidences of Adverse Events in Patients Excluded from the Safety Analysis Set

Analysis set: Patients excluded from the Safety Analysis Set

Data element AEs

analyzed:

Analysis method: The above-mentioned data element will be analyzed using the same method

described in section 4.1.1.

#### 4.2.2 Incidences of Adverse Drug Reactions/Infections in Patients Excluded from the Safety **Analysis Set**

Analysis set: Patients excluded from the Safety Analysis Set

Data element ADRs, etc.

analyzed:

Analysis method: The above-mentioned data element will be analyzed using the same method

described in section 4.1.2.

#### Incidences of Adverse Events and Adverse Drug Reactions/Infections by Seriousness, 4.3 Time of Onset, Outcome, and Causal Relationship with Fomepizole IV

#### 4.3.1 Incidences of Adverse Events by Seriousness, Time of Onset, Outcome, and Causal Relationship with Fomepizole IV

Analysis set: Safety Analysis Set

Data element **AEs** 

analyzed:

Stratification Total

variable:

Seriousness

[Min <= - < 24, 24 <= - < 48, 48 <= - < Time of onset (time)

Outcome [recovered/resolved, recovering/resolving,

not recovered/not resolved,

recovered/resolved with sequelae, death

(due to this event), unknown]

Causal relationship to fomepizole [related, not related]

Property of Lakeda Analysis method: The above-mentioned data elements will be analyzed using the same method described in section 4.1.1 for each stratum of the stratification variables. Patients

with multiple occurrences of the same SOC/PT will be counted as a single patient within said SOC/PT. Events in the same SOC will be analyzed as single

events according to the priority described below, whereas events with the same

PT will be analyzed as single events according to the priority described below

based on the details of the stratification variable.

Seriousness: Serious→Not serious

Time of onset:  $<24 \text{ hr} \rightarrow 24 \text{-} <48 \text{ hr} \rightarrow 48 \text{-} <72 \text{ hr} \rightarrow 72 \text{-} <96 \text{ hr} \rightarrow 96 \text{-} <120 \text{ hr} \rightarrow$ 

≥120 hr

Outcome: Death (due to this event)  $\rightarrow$  Recovered/resolved with sequelae  $\rightarrow$  Not recovered/not resolved  $\rightarrow$  Recovering/resolving  $\rightarrow$  Recovered/resolved  $\rightarrow$ 

Unknown

Causal relationship with fomepizole IV: Related→ Not related

#### 4.3.2 Incidences of Adverse Drug Reactions/Infections By Seriousness, Time of Onset, and Outcome

Analysis set: Safety Analysis Set

Data element ADRs, etc.

analyzed:

Stratification Total

variable:

[serious, not serious] Seriousness

Time of onset (time)

 $\leq Max$ 

Outcome recovered/resolved, recovering/resolving,

not recovered/not resolved,

recovered/resolved with sequelae, death

(due to this event), unknown]

The above-mentioned data elements will be analyzed using the same method Analysis method:

described in section 4.1.2 for each stratum of the stratification variables. Patients

with multiple occurrences of the same SOC/PT will be counted as a single

patient within said SOC/PT. Events in the same SOC will be analyzed as single

events according to the priority described below, whereas events with the same

PT will be analyzed as single events according to the priority described below

based on the details of the stratification variable.

Seriousness: Serious→Not serious

Time of onset:  $<24 \text{ hr} \rightarrow 24 < 48 \text{ hr} \rightarrow 48 < 72 \text{ hr} \rightarrow 72 < 96 \text{ hr} \rightarrow 96 < 120 \text{ hr} \rightarrow$ 

≥120 hr

Outcome: Death (due to this event) → Recovered/resolved with sequelae → Not

recovered/not resolved → Recovering/resolving → Recovered/resolved →

Unknown

# Property of Lakedai. For Incidences of Serious Adverse Events and Adverse Drug Reactions/Infections

#### 4.4.1 Incidences of Serious Adverse Events

Analysis set: Safety Analysis Set Data element **SAEs** 

analyzed:

Analysis method:

#### 4.4.2 Incidences of Serious Adverse Drug Reactions/Infections

Analysis set: Data element

analyzed:

Analysis method:

#### **Factors Potentially Affecting Safety**

# The above-mentioned data element will be analyzed using the same method described in section 4.1.2. ially Affecting Safety Adverse Drug Reactions/Inferrage and Treatment Property of Takeda. For noncommercial use only and subject to the property of Takeda. 4.5.1 Incidences of Adverse Drug Reactions/Infections by Patient Demographics & Baseline

 $[Min \le - < 65, 65 \le - < = Max,]$ 

Unknown]

[male, female]

[Min <= - < 65, 65 <= - <= 74, 75 <=

- <= Max, Unknown]

 $[Min \le - < 20, 20 \le - < 29, 30 \le -$ 

- <= 39, 40 <= - <= 49, 50 <= - <=

 $59, 60 \le - \le 69, 70 \le - \le 79,$ 

 $80 \le - \le Max$ , Unknown

[no, yes, unknown]

[15 mg/kg, 10 mg/kg, Other]

[no, yes]

[no, yes]

[no, yes]

[no, yes]

than fomepizole IV)

Toxic symptoms (at start of fomepizole [no, yes]

IV dosing)

The above-mentioned data elements will be analyzed for each stratum of the Analysis method: stratification variables as follows.

- No. of patients with ADRs, etc. (1)
- (2) No. of occurrences of ADRs, etc.
- Incidence rate of ADRs, etc. (3)

Each of these data elements will be determined as follows.

No. of patients with ADRs, etc.:

The number of patients who develop ADRs, etc.

Number of occurrences of ADRs, etc.:

The number of times that ADRS, etc. occur.

Incidence rate of ADRs, etc.:

Calculated as follows: No. of patients with ADRs, etc. ÷ No. of patients in the Safety Analysis Set × 100

#### 4.5.2 Incidences of Adverse Drug Reactions/Infections by Seriousness, Deaths, Patient **Demographics & Baseline Characteristics and Treatment Details**

Analysis set:

Data element

analyzed:

Stratification [serious, not serious]

variable 1:

Property of Takedai. For not A Stratification [male, female]

Age (years)  $Min \le -65, 65 \le - \le Max$ 

Unknown]

 $Min \le -65, 65 \le -874, 75 \le$ 

- <= Max, Unknown]

[no, yes, unknown]

 $Min \le -20, 20 \le -29, 30 \le$ 

- <= 39, 40 <= - <= 49, 50 <= - <=

 $59, 60 \le - \le 69, 70 \le - \le 79,$ 

 $80 \le - \le \text{Max}, \text{Unknown}$ 

Alcohol consumption (at time of

poisoning)

Infusion dose per body weight [15 mg/kg, 10 mg/kg, Other] Acute blood purification therapy [no, yes]

Respiratory management (mechanical [no, yes]

ventilation)

GI decontamination [no, yes]

Administration of medication (other [no, yes]

than fomepizole IV)

Toxic symptoms (at start of fomepizole [no, yes]

IV dosing)

Analysis method: The dual stratification variables 1 and 2 for the above-mentioned data elements

will be analyzed using the same method described in section 4.5.1.

#### 4.5.3 Incidences of Adverse Drug Reactions/Infections by Sex

Analysis set: Safety Analysis Set

Data element ADRs, etc.

analyzed:

Stratification Sex [male, female

variable:

Analysis method: The above-mentioned data elements will be analyzed using the same method

described in section 4.1.2 for each stratum of the stratification variables.

#### 4.5.4 Incidences of Adverse Drug Reactions/Infections by Age Bracket

Analysis set: Safety Analysis Set

Data element ADRs, etc.

analyzed:

Stratification Age (years)  $[Min \le - < 65, 65 \le - \le - \le Max, Unknown]$ 

variable:  $[Min \le - < 65, 65 \le - < 74, 75 \le - < Max,]$ 

Unknown]

[Min <= - < 20, 20 <= - <= 29, 30 <= - <= 39, 40 <= - <=

49, 50 <= - <= 59, 60 <= - <= 69, 70 <= - <= 79, 80 <=

- <= Max, Unknown]

Analysis method: The above-mentioned data elements will be analyzed using the same method

described in section 4.1.2 for each stratum of the stratification variables.

#### 4.5.5 Incidences of Adverse Drug Reactions/Infections by Alcohol Consumption (Y/N)

Analysis set: Safety Analysis Set

Data element ADRs, etc.

analyzed:

Stratification Alcohol consumption (at time of [no, yes, unknown]

variable: poisoning)

Analysis method: The above-mentioned data elements will be analyzed using the same method

described in section 4.1.2 for each stratum of the stratification variables.

#### 4.5.6 Incidences of Adverse Drug Reactions/Infections by Administration of Fomepizole IV

Analysis set: Safety Analysis Set

Data element ADRs, etc.

analyzed:

Stratification Infusion dose per body weight [15 mg/kg, 10 mg/kg, Other]

variable:

Analysis method: The above-mentioned data elements will be analyzed using the same method

described in section 4.1.2 for each stratum of the stratification variables.

## 4.5.7 Incidences of Adverse Drug Reactions/Infections by Intervention/Procedure (Other than Pharmacotherapy)

Analysis set: Safety Analysis Set

Data element ADRs, etc.

analyzed:

Stratification Acute blood purification therapy [no, yes]

variable:

Respiratory management (mechanical [no, yes]

ventilation) 0

GI decontamination [no, yes]

Analysis method: The above-mentioned data elements will be analyzed using the same method

described in section 4.1.2 for each stratum of the stratification variables.

## 4.5.8 Incidences of Adverse Drug Reactions/Infections by Administration of Medications (Other than Fomepizole IV)

Analysis set: Safety Analysis Set

Data element ADRs, etc.

analyzed:

Stratification Administration of medication [no, yes]

variable: (other than fomepizole IV)

Analysis method: The above-mentioned data elements will be analyzed using the same method

described in section 4.1.2 for each stratum of the stratification variables.

#### 4.5.9 Incidences of Adverse Drug Reactions/Infections by Presence or Absence (Y/N) of Toxic **Symptoms**

Analysis set: Safety Analysis Set

Data element ADRs, etc.

analyzed:

Stratification Toxic symptoms [no, yes]

variable:

Analysis method: The above-mentioned data elements will be analyzed using the same method

described in section 4.1.2 for each stratum of the stratification variables.

#### **Time Courses of Test and Measurement Data** 4.6

#### 4.6.1 Time Courses of Vital Signs

Analysis set: Safety Analysis Set

Pulse rate, systolic blood pressure, diastolic blood pressure, respiratory rate, Data element

analyzed: body temperature

At start of fomepizole IV dosing (i.e., baseline), 0.5 hr after start of fomepizole Assessment IV dosing, 4 hr after start of fomepizole IV dosing, 8 hr after start of fomepizole timepoints:

IV dosing, 12 hr after start of fomepizole IV dosing, 16 hr after start of

fomepizole IV dosing, 20 hr after start of fomepizole IV dosing, 24 hr after start of fomepizole IV dosing, 36 hr after start of fomepizole IV dosing, 48 hr after start of fomepizole IV dosing, 60 hr after start of fomepizole IV dosing, 72 hr after start of fomepizole IV dosing, 84 hr after start of fomepizole IV dosing, 96 hr after start of fomepizole IV dosing, 108 hr after start of fomepizole IV dosing, at completion of final fomepizole IV infusion, 12 hr after completion of final fomepizole IV infusion, 24 hr after completion of final fomepizole IV infusion,

at final assessment

Analysis method: Summary statistics of the above-mentioned data elements will be presented for

> measured values and absolute changes from baseline (obtained by subtracting the measured values at the start of fomepizole IV dosing [i.e., at baseline] from the measured value at each assessment timepoint after starting fomepizole IV dosing), and the 95% CI of the mean will be presented for said absolute changes

> from baseline. Spaghetti graphs will also be prepared for the measured values of

all patients.

## Property of Lakedia. 4.6.2 Time Courses of Laboratory Test Parameters

Analysis set: Safety Analysis Set Data element RBC count, WBC count, platelet count, AST, ALT, gamma-GTP, serum

analyzed: creatinine, BUN

At start of fomepizole IV dosing (i.e., baseline), 0.5 hr after start of fomepizole Assessment

IV dosing, 4 hr after start of fomepizole IV dosing, 8 hr after start of fomepizole timepoints:

IV dosing, 12 hr after start of fomepizole IV dosing, 16 hr after start of

fomepizole IV dosing, 20 hr after start of fomepizole IV dosing, 24 hr after start of fomepizole IV dosing, 36 hr after start of fomepizole IV dosing, 48 hr after start of fomepizole IV dosing, 60 hr after start of fomepizole IV dosing, 72 hr after start of fomepizole IV dosing, 84 hr after start of fomepizole IV dosing, 96 hr after start of fomepizole IV dosing, 108 hr after start of fomepizole IV dosing, at completion of final fomepizole IV infusion, 12 hr after completion of final fomepizole IV infusion, 24 hr after completion of final fomepizole IV infusion,

at final assessment

Summary statistics of the above-mentioned data elements will be presented for Analysis method:

> test values and absolute changes from baseline (obtained by subtracting the test values at the start of fomepizole IV dosing [i.e., at baseline] from the test value at each assessment timepoint after starting fomepizole IV dosing), and the 95%

pres. All also by the property of Takeda. For non-commercial use CI of the mean will be presented for said absolute changes from baseline.

Spaghetti graphs will also be prepared for the test values of all patients.

#### 5 EFFICACY ANALYSES

#### 5.1 Time Course of Arterial Blood pH

Analysis set: Patients in the Efficacy Analysis Set for whom test value/s from at least one

assessment time point is/are available from both before (i.e., at baseline) and

after the start of fomepizole IV dosing.

Data element Arterial blood gas analysis (arterial blood pH)

analyzed:

Assessment At start of fomepizole IV dosing (i.e., baseline), 0.5 hr after start of fomepizole

timepoints: IV dosing, 4 hr after start of fomepizole IV dosing, 8 hr after start of fomepizole

IV dosing, 12 hr after start of fomepizole IV dosing, 16 hr after start of

fomepizole IV dosing, 20 hr after start of fomepizole IV dosing, 24 hr after start of fomepizole IV dosing, 36 hr after start of fomepizole IV dosing, 48 hr after start of fomepizole IV dosing, 60 hr after start of fomepizole IV dosing, 72 hr after start of fomepizole IV dosing, 84 hr after start of fomepizole IV dosing, 96 hr after start of fomepizole IV dosing, 108 hr after start of fomepizole IV dosing, at completion of final fomepizole IV infusion, 12 hr after completion of final fomepizole IV infusion,

at final assessment

Analysis method: Summary statistics of the above-mentioned data elements will be presented for

test values and absolute changes from baseline (obtained by subtracting the test values at the start of fomepizole IV dosing [i.e., at baseline] from the test value at each assessment timepoint after starting fomepizole IV dosing). The 95% CI

of the mean will also be presented and a paired Student's t-test will be

performed for absolute changes from baseline. Furthermore, line graphs will be prepared by plotting the mean±SD of test values on the Y-axis and the test

timepoints on the X-axis, while bar graphs will be prepared by plotting

absolute changes from baseline on the Y-axis and the test timepoints on the

X-axis. The results of the paired Student's t-test will be denoted within the

graph with an asterisk (\*).

#### 5.2 Time Courses of Poisoning/Toxicity Test Parameters

Analysis set: Patients in the Efficacy Analysis Set for whom test value/s from at least one

assessment time point is/are available from both before (i.e., at baseline) and

after the start of fomepizole IV dosing.

Data element Arterial blood gas analyses (arterial carbon dioxide partial pressure [PaCO<sub>2</sub>],

analyzed: arterial oxygen partial pressure [PaO<sub>2</sub>], bicarbonate ion, base excess [BE], anion

gap, blood ethylene glycol concentration, blood glycolic acid concentration, blood methanol concentration, blood formic acid concentration, osmotic pressure gap)

Assessment timepoints:

At start of fomepizole IV dosing (i.e., baseline), 0.5 hr after start of fomepizole IV dosing, 4 hr after start of fomepizole IV dosing, 8 hr after start of fomepizole IV dosing, 12 hr after start of fomepizole IV dosing, 16 hr after start of fomepizole IV dosing, 20 hr after start of fomepizole IV dosing, 24 hr after start of fomepizole IV dosing, 36 hr after start of fomepizole IV dosing, 48 hr after start of fomepizole IV dosing, 60 hr after start of fomepizole IV dosing, 72 hr after start of fomepizole IV dosing, 84 hr after start of fomepizole IV dosing, 96 hr after start of fomepizole IV dosing, 108 hr after start of fomepizole IV dosing, at completion of final fomepizole IV infusion, 12 hr after completion of final fomepizole IV infusion, at final assessment

Analysis method:

Summary statistics of the above-mentioned data elements will be presented for test values and absolute changes from baseline (obtained by subtracting the test values at the start of fomepizole IV dosing [i.e., at baseline] from the test value at each assessment timepoint after starting fomepizole IV dosing). The 95% CI of the mean will also be presented and a paired Student's t-test will be performed for absolute changes from baseline. Furthermore, line graphs will be prepared by plotting the mean±SD of test values on the Y-axis and the test timepoints on the X-axis, while bar graphs will be prepared by plotting absolute changes from baseline on the Y-axis and the test timepoints on the X-axis. The results of the paired Student's t-test will be denoted within the graph with an asterisk (\*).

#### 5.3 Time Courses of Toxic Symptoms

Analysis set: Patients in the Efficacy Analysis Set for whom data is available for at least one

toxic symptom parameter both at baseline and at completion of the final

fomepizole IV infusion.

Data element

analyzed:

Respiratory symptoms (tachypnea, respiratory failure, laboured breathing)

Cardiovascular symptoms (cardiovascular irritation, tachycardia, bradycardia,

arrhythmias, hypertension, heart failure)

GI symptoms (nausea, vomiting, abdominal pain)

Neurologic or psychiatric symptoms (nervous system irritation, consciousness

disturbed, convulsions, ataxia)

Renal and urinary symptoms (renal failure, hematuria)

Eye symptoms (visual impairment, nystagmus)

Abnormal test values (renal function test abnormal, liver function test abnormal, electrolytes abnormal (sodium abnormal, potassium abnormal, calcium abnormal, phosphorus abnormal, magnesium abnormal), metabolic acidosis (examination finding), urine sediment abnormal, osmotic pressure gap abnormal, chest X-ray abnormal, electrocardiography abnormal, cranial CT

abnormal, brain edema on MRI, fundus examination abnormal).

Assessment At the start of fomepizole IV dosing (i.e., at baseline) and at completion of the

timepoints: final fomepizole IV infusion

Analysis method: The numbers and proportions of patients with or without each toxic symptom at

each assessment timepoint will be presented for each of the above-mentioned data elements. Presence or absence of toxic symptoms at baseline will also be cross-tabulated against those at completion of the final fomepizole IV infusion.

5.4 Outcome

Analysis set: Patients in the Efficacy Analysis Set and patients in the Safety Analysis Set for

whom outcome was recorded in the CRF.

Data element Outcome [survived without sequelae, survived

analyzed: with sequelae, death]

Sequelae details

\* Only if the outcome is "survived

with sequelae"

Analysis method: Frequency tables will be prepared for each outcome in the above-mentioned data

elements in both the Efficacy Analysis Set and in the Safety Analysis Set.

Listings will also be prepared for the Safety Analysis Set and Efficacy Analysis

Set categories, outcomes and details of sequelae.

5.5 Factors Potentially Affecting Efficacy

Analysis set: Patients in the Efficacy Analysis Set for whom test value/s from at least one

assessment time point is/are available from both before (i.e., at baseline) and

after the start of fomepizole IV dosing.

Data element Arterial blood gas analysis (arterial blood pH)

analyzed:

Assessment At start of fomepizole IV dosing (i.e., baseline), 0.5 hr after start of fomepizole

timepoints: IV dosing, 4 hr after start of fomepizole IV dosing, 8 hr after start of fomepizole

IV dosing, 12 hr after start of fomepizole IV dosing, 16 hr after start of fomepizole IV dosing, 20 hr after start of fomepizole IV dosing, 24 hr after start of fomepizole IV dosing, 36 hr after start of fomepizole IV dosing, 48 hr after start of fomepizole IV dosing, 60 hr after start of fomepizole IV dosing, 72 hr after start of fomepizole IV dosing, 84 hr after start of fomepizole IV dosing, 96 hr after start of fomepizole IV dosing, 108 hr after start of fomepizole IV dosing, at completion of final fomepizole IV infusion, 12 hr after completion of final fomepizole IV infusion, 24 hr after completion of final fomepizole IV infusion, at final assessment

Stratification

Sex [male, female]

variable:

[Min <= - < 65, 65 <= Max, Age (years)

[Min <= - < 65, 65 <= - <= 74, 75 <= - <= Max, Unknown]

[Min <= - < 20, 20 <= - <= 29, 30 <= - <= 39, 40 <= - <= 49, 50 <= - <= 59, 60 <= - <= 69, 70 <= - <= 79, 80 <= - <= Max,

Unknown]

Alcohol consumption (at time of

[no, yes, unknown]

poisoning)

Infusion dose per body weight [15 mg/kg, 10 mg/kg, Other]

Acute blood purification therapy [no, yes] Respiratory management [no, yes]

(mechanical ventilation)

GI decontamination [no, yes]

Administration of medication [no, yes]

(other than fomepizole IV)

Toxic symptoms [no, yes]

Summary statistics for test values at each assessment timepoint will be calculated for each stratum of the stratification variable of the data elements listed above.

#### INCIDENCE OF ADVERSE DRUG REACTIONS/INFECTIONS IN THE SUPPLEMENTARY PHARMACOVIGILANCE PLAN

#### 6.1 Incidence of Adverse Drug Reactions/Infections in the Supplementary Pharmacovigilance Plan (Attached Form 12)

Analysis set: Safety Analysis Set

Data element ADRs, etc. in the Safety Specification (important identified risks, important

analyzed: potential risks, and important missing information)

Stratification [serious, not serious] Seriousness

variable:

Analysis of the above-mentioned data elements will be performed for each Analysis

method: stratum of the stratification variables as follows according to Attached Form 12

(Notes) items 1 through 4 stipulated in Re-Examination Notification No. 0325-10

issued on 25 March 2020 by the Pharmaceutical Evaluation Division,

Pharmaceutical Safety and Environmental Health Bureau, Ministry of Health,

Labour and Welfare (herein "MHLW/PSEHB/PED").

Numbers and incidence rates of patients with ADRs, etc.

The names of risks and the order of describing these risks shall adhere to the sing Info.
sing Info.
sing Info.
property of Lakeda. For non-commercial use definitions outlined in the Important Identified Risks, Important Potential Risks,

and Important Missing Information.

#### SUMMARY OF PATIENTS IN POSTMARKETING SURVEILLANCE

# 3ct to the applicable reins of Use **Summary of Patients in Postmarketing Surveillance (Attached Form 16)** 7.1

Analysis set: Patients for whom CRFs were submitted/collected

Data element Patient No.

analyzed:

Site name

Sex

Age

Reason for use (disease code, disease name)

Concomitant disease (disease code, disease name)

Route of administration

Maximum dose

Mean dose

Units

Period used (duration of fomepizole IV treatment)

Concomitant medications (drug code, drug name)

Extent of response

ADRs (disease code, disease name, outcome)

CRF number

Dropouts

Reason for dropout

Listings of the above-mentioned data elements will be prepared in accordance Analysis

Jf the "Proce MHLWPSEHB, November 2020. with the "Procedures for Preparing Reexamination Data Entry Files" stipulated in

MHLW/PSEHB/PEB Re-Examination Notification No. 1119-3 issued on 19

#### **Document History (Version Control)**

| | Version Original | Date 2015.10.23 | Created or modified by | Comments New document |
|---|---|---|---|---|
| | version 2nd version | 2022.6.23 | | The tabulated data was revised in accordance with the SAP standardized template. |
| | Version 2.1 | 2022.8.1 | | Version 2.1 created All changes from Version 2 are described in Attachment 1. |
| Property | akeda | Fornonic | ommercialue | Version 2.1 created All changes from Version 2 are described in Attachment 1. |

35

#### [Attachment 1] Amendment Comparison Table

Statistical Analysis Plan (Version 2: Prepared on 23 June 2022 → Version 2.1: Prepared on 1 August 2022)

| Statistical 1 III | arysis riam (version 2: rrepared on 25 vane 2022 | version 2:1: 11eparea on 111agust 2022) | 110 |
|---|---|---|---|
| Page No. | Before amendment | After amendment | Reason for amendment |
| 13 | Description of level of consciousness | Description of level of consciousness | Due to a change in the method of analysis, the |
| | assessment: | assessment: | 3-3-9 rating system (JCS) category "0 (alert)" |
| | 3-3-9 rating system (JCS): [I, II, III] | 3-3-9 rating system (JCS): [0 (alert), I, II, III] | was added to the analyzed data element "Level |
| | | sie | of consciousness details" in section 2.1 |
| | | END, | "Patient Demographics and Baseline |
| | | .03 | Characteristics." |
| | | 3 | |
| | | and a second | |